CLINICAL TRIAL: NCT04319120
Title: Pilot Study of descriPtion of cicatriSation Rates of Digital Ulcers in Systemic scleroDerma
Acronym: POPSUD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI18_0017
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Scleroderma, Systemic
Keywords: Scleroderma - Digital Ulcers
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- questionnaires online: Each month, the nurse will contact the patients included, by mail or telephone, to fill out their questionnaires online or by mail, and to make a photo of the ulcer if it is healed.
  Interventions: Other: questionnaires online

INTERVENTIONS:
Other: questionnaires online — Each month, the nurse will contact the patients included, by mail or telephone, to fill out their questionnaires online or by mail, and to make a photo of the ulcer if it is healed. A dedicated telephone line and e-mail address will be used as a support if necessary (for questionnaires, emails or sending photos). The referring nurse and the clinical research assistant of the service will be in charge of centralizing the data collected.

SUMMARY:
To make an updated inventory of digital ulcer care protocols in scleroderma patients and to specify the French data on monthly healing rates and local care with patients in care centers experience, and thus to know the impact of ulcers in different dimensions To evaluate the rate of healed digital ulcers at the end of the study

ELIGIBILITY:
Inclusion Criteria:

* Patient with systemic scleroderma according to the ACR / EULAR 2012 criteria
* Patient with one or more active digital ulcers
* Patient with internet access and camera or smartphone

Exclusion Criteria:

* Minor patients
* Patient deprived of liberty or subject to a court order
* Patient subject to a legal protection measure
* Pregnant or lactating woman
* Patient unable to complete the questionnaires

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with systemic scleroderma
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of digital ulcers | 1 year
  Number of digital ulcers healed at the end of the study

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Bordeaux Hospital, Bordeaux
  - Limoges Hospital, Limoges
  - Toulouse Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No